CLINICAL TRIAL: NCT04351464
Title: Is Reflexology Applied to Children With Cerebral Palsy an Effective Method?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Sabiha BEZGİN, PhD, Physical Therapist, Kırıkkale University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: SBEZGIN
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Cerebral Palsy; Reflexology
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy and Reflexology group (Active Comparator): Received reflexology implementation for 20-30 minutes on the sole along with the physical treatment involving NDT approaches. Within the scope of the implementation, all the reflex points on the sole were stimulated. The pituitary gland, which is related to sleep and control of salivation, oromotor area and areas of muscular and skeletal system were stimulated with further repetitions.
  Interventions: Other: physical therapy and reflexology
- Just Physical therapy group (Experimental): The group received a 45-minute physical therapy program involving NDT approaches as the control group. Within the scope of this program, the children were treated with intramuscular stretching and soft tissue mobilization, exercises that improved balance and that supported the development of postural control, position shifts, and stretching and reinforcement exercises in the necessary muscle groups.
  Interventions: Other: physical therapy and reflexology

INTERVENTIONS:
Other: physical therapy and reflexology

SUMMARY:
Objectives: This study was planned to investigate the influence of reflexology applied to children with cerebral palsy together with physical therapy program involving neurodevelopmental approaches.

Methods: The study involved 40 children aged,16 girls and 24 boys between 3 and 15 years and divided into two groups. While the children in Group 1 were given twice a week for eight weeks neurodevelopmental treatment, reflexology was applied to those in Group 2 together with neurodevelopmental treatment. Drooling Severity and Frequency Scale, Pediatric Sleep Questionnaire and the Children's Health Questionnaire was used to assess the drooling, status of sleep and quality of life in children.

DETAILED DESCRIPTION:
The study involved a total of 40 children aged between three and 15 diagnosed with CP by a pediatric neurologist. Children at levels 3/4/5 of the GMFCS who did not have any open wounds on the foot, where the application was to be performed, and whose parents consented to the child's participation were accepted in the study. However, those children were excluded who were treated with botulinum toxin in the last six months, underwent surgery, were treated with reflexology or any other alternative medicine method and who had refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Children at levels 3/4/5 of the GMFCS who did not have any open wounds on the foot, where the application was to be performed, and whose parents consented to the child's participation were accepted in the study.

Exclusion Criteria:

* who were treated with botulinum toxin in the last six months, underwent surgery, were treated with reflexology or any other alternative medicine method and who had refractory epilepsy.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
physiological parameter | 8 weeks
  Drooling frequency and severity of drooling
Questionnaire about Sleep status | 8 weeks
  Assess the problems related to sleep
Questionnaire about Quality of life of children | 8 weeks
  general health, physical condition, global behavior, mental health, self-esteem and the effect of time on parents

SECONDARY OUTCOMES:
Physical parameter | 8 weeks
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Sabiha Bezgin, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided